CLINICAL TRIAL: NCT02267395
Title: Scapular and Cervical Neuromuscular Deficits in Musicians With and Without Playing Related Musculoskeletal Disorders: A Case Control Study.
Brief Title: Scapular and Cervical Neuromuscular Control Deficits in Musicians With and Without Playing Injuries.
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Flavio Silva, Clinical Coordinator of Physical Therapy, Vanderbilt University
Other Study IDs: 1212
Record Dates: First submitted 2014-09-29; First posted 2014-10-17 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Playing Related Musculoskeletal Disorders
Keywords: Musicians, Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- (No-PRMSDs): Group 1 : No Playing Related Musculoskeletal Injury
  Interventions: Other: (1) cranio-cervical flexion test;; Other: (2) scapular dyskinesis test; Other: (3) deep neck flexor endurance test.
- (Yes-PRMSDs): Group 2: Playing Related Musculoskeletal Injury
  Interventions: Other: (1) cranio-cervical flexion test;; Other: (2) scapular dyskinesis test; Other: (3) deep neck flexor endurance test.

INTERVENTIONS:
Other: (1) cranio-cervical flexion test; — Test to determine level of strength for Deep Neck Flexor muscles
Other: (2) scapular dyskinesis test — Test to determine scapular control
Other: (3) deep neck flexor endurance test. — Test do determine endurance for the deep neck flexor muscle group.

SUMMARY:
The study will investigate if there are differences in the presence of: (1) prior injury, playing patterns, and physical fitness habits; (2) scapular control; and (3) cervical neuromuscular control and endurance deficits between musicians with and without current playing related musculoskeletal injuries.

DETAILED DESCRIPTION:
Background: The art of professionally playing a musical instrument can be physically demanding. Such activity involves maintaining static postures and producing repetitive motions for countless hours of playing time between practice and performances, often with very little rest. More than 50% of musicians will develop upper extremity injuries and pain related to instrument use, which can negatively affect or interrupt their careers. Efficient cervical spine and shoulder girdle neuromuscular control is essential for upper quarter musculoskeletal injury prevention. Neuromuscular control deficits are linked to a higher upper extremity occupational injury incidence in most professions. However, no research to date has investigated if there are differences in scapular and cervical endurance and neuromuscular control between musicians with and without playing-related cervical and upper extremity musculoskeletal disorders.

Design: Case-control study Setting: Musical venue and university setting. Participants: Eighty subjects including student musicians from different universities and professional musicians in Tennessee.

Methods: Musicians will be consecutively recruited to fill in a questionnaire regarding the presence of cervical and upper extremity PRMSDs. Those subjects with PRMSDs (Yes-PRMSDs) will undergo clinical testing for the presence of scapular dyskinesis and cervical neuromuscular control and endurance deficits using the following tests: (1) cranio-cervical flexion test; (2) scapular dyskinesis test; and (3) deep neck flexor endurance test. Asymptomatic musicians (No-PRMSDs) will be recruited consecutively, matched by gender, type of instrument (string instrument or other) and number of hours played per week and tested following the same protocol.

Reliability testing: To determine intrarater reliability prior to data collection, a convenience sample of twenty subjects not included in the study will be evaluated over two days for (1) Cranio-cervical flexion test; (2) Scapular dyskinesis test; and (3) deep neck flexor endurance test. Tests will be repeated with at least a 24-hour interval between testing sessions. Intra-class correlation coefficient (model 3, 2) for the two cervical tests and Kappa statistics model for the scapular dyskinesis test will be calculated for determination of intrarater reliability.

Interventions: Subjects will complete a comprehensive demographic questionnaire that includes playing patterns, as well as general health related questions and fitness activities exposure. In a second visit, subjects in both groups will complete a test battery that includes cranio-cervical flexion test, scapular dyskinesis assessment and deep neck flexor endurance test. Blinding of the assessor as to the group in which subjects are members (Yes-PRMSDs versus No-PRMSDs) will be ensured.

Purpose: The purposes of this research will be to investigate if there are differences in the presence of: (1) prior injury, playing patterns, and physical fitness habits; (2) scapular dyskinesis; and (3) cervical neuromuscular control and endurance deficits between musicians with and without playing related musculoskeletal Disorders (PRMSDs)

ELIGIBILITY:
Inclusion Criteria for Experimental Group:

1. Student musicians or professional musicians playing instrument 6 hours or more per week.
2. Current pain or history of cervical or upper extremity PRMSDs and or history of pain during the past year with symptoms lasting more than one week and affecting musical performance.
3. Between 18 and 65 years of age.

Inclusion Criteria for Control group:

1. Student musician or professional musician playing instrument more than 6 hours a week.
2. No history of cervical or upper extremity injury and or pain during the past year with symptoms lasting more than one week
3. Between 18 and 65 years of age.

Exclusion Criteria:

1. History of trauma or injury other than playing related injury, currently affecting the ability to play musical instrument.
2. Pregnancy
3. Neurological disorder affecting motor control (including but not limited to Parkinson' s, multiple sclerosis, Amyotrophic lateral sclerosis, muscular dystrophy, myasthenia gravis, Guillain-Barre)
4. Rheumatoid arthritis or ankylosing spondylitis
5. Diagnosis of any connective tissue disorder (Including but not limited to Marfan's syndrome, Ehlers-Danlos syndrome, systemic lupus erythematosus, scleroderma)
6. Presence of cervical radiculopathy
7. History of recent (within the last year) cervical or shoulder surgery

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Musicians with and without playing related musculo-skeletal Injuries.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cranio Cervical Flexion test Score | 1 day
  Score of Cranio Cervical Flexion test
Presence of scapular dyskinesia | 1
  Presence of scapular dyskinesia
Deep Neck Flexor Endurance Test Score | 1
  Score of Deep Neck Flexor Endurance test

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Silva, BscPT, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Orthopaedics Cool Springs, Franklin, Tennessee, United States

REFERENCES:
- [Background] Ackermann B, Driscoll T, Kenny DT. Musculoskeletal pain and injury in professional orchestral musicians in Australia. Med Probl Perform Art. 2012 Dec;27(4):181-7. PMID 23247873
- [Background] Barton PM, Hayes KC. Neck flexor muscle strength, efficiency, and relaxation times in normal subjects and subjects with unilateral neck pain and headache. Arch Phys Med Rehabil. 1996 Jul;77(7):680-7. doi: 10.1016/s0003-9993(96)90008-8. PMID 8669995
- [Background] Bruno S, Lorusso A, L'Abbate N. Playing-related disabling musculoskeletal disorders in young and adult classical piano students. Int Arch Occup Environ Health. 2008 Jul;81(7):855-60. doi: 10.1007/s00420-007-0279-8. Epub 2008 Jan 22. PMID 18210148
- [Background] Chan C, Driscoll T, Ackermann B. Development of a specific exercise programme for professional orchestral musicians. Inj Prev. 2013 Aug;19(4):257-63. doi: 10.1136/injuryprev-2012-040608. Epub 2012 Dec 4. PMID 23211353
- [Background] Chiu TT, Law EY, Chiu TH. Performance of the craniocervical flexion test in subjects with and without chronic neck pain. J Orthop Sports Phys Ther. 2005 Sep;35(9):567-71. doi: 10.2519/jospt.2005.35.9.567. PMID 16268243
- [Background] Cools AM, Struyf F, De Mey K, Maenhout A, Castelein B, Cagnie B. Rehabilitation of scapular dyskinesis: from the office worker to the elite overhead athlete. Br J Sports Med. 2014 Apr;48(8):692-7. doi: 10.1136/bjsports-2013-092148. Epub 2013 May 18. PMID 23687006
- [Background] De Mey K, Danneels L, Cagnie B, Cools AM. Scapular muscle rehabilitation exercises in overhead athletes with impingement symptoms: effect of a 6-week training program on muscle recruitment and functional outcome. Am J Sports Med. 2012 Aug;40(8):1906-15. doi: 10.1177/0363546512453297. Epub 2012 Jul 11. PMID 22785606
- [Background] Dick RW, Berning JR, Dawson W, Ginsburg RD, Miller C, Shybut GT. Athletes and the arts--the role of sports medicine in the performing arts. Curr Sports Med Rep. 2013 Nov-Dec;12(6):397-403. doi: 10.1249/JSR.0000000000000009. PMID 24225525
- [Background] Domenech MA, Sizer PS, Dedrick GS, McGalliard MK, Brismee JM. The deep neck flexor endurance test: normative data scores in healthy adults. PM R. 2011 Feb;3(2):105-10. doi: 10.1016/j.pmrj.2010.10.023. PMID 21333948
- [Background] Falla D, O'Leary S, Farina D, Jull G. The change in deep cervical flexor activity after training is associated with the degree of pain reduction in patients with chronic neck pain. Clin J Pain. 2012 Sep;28(7):628-34. doi: 10.1097/AJP.0b013e31823e9378. PMID 22156825
- [Background] Fry HJ. Overuse syndromes in instrumental musicians. Semin Neurol. 1989 Jun;9(2):136-45. doi: 10.1055/s-2008-1041317. No abstract available. PMID 2557662
- [Background] Grieco A, Occhipinti E, Colombini D, Menoni O, Bulgheroni M, Frigo C, Boccardi S. Muscular effort and musculo-skeletal disorders in piano students: electromyographic, clinical and preventive aspects. Ergonomics. 1989 Jul;32(7):697-716. doi: 10.1080/00140138908966837. PMID 2806217
- [Background] Harris KD, Heer DM, Roy TC, Santos DM, Whitman JM, Wainner RS. Reliability of a measurement of neck flexor muscle endurance. Phys Ther. 2005 Dec;85(12):1349-55. PMID 16305273
- [Background] Hidalgo-Lozano A, Calderon-Soto C, Domingo-Camara A, Fernandez-de-Las-Penas C, Madeleine P, Arroyo-Morales M. Elite swimmers with unilateral shoulder pain demonstrate altered pattern of cervical muscle activation during a functional upper-limb task. J Orthop Sports Phys Ther. 2012 Jun;42(6):552-8. doi: 10.2519/jospt.2012.3875. Epub 2012 Jan 25. PMID 22282107
- [Background] Holmgren T, Bjornsson Hallgren H, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. BMJ. 2012 Feb 20;344:e787. doi: 10.1136/bmj.e787. PMID 22349588
- [Background] Hoppmann RA. Instrumental musicians' hazards. Occup Med. 2001 Oct-Dec;16(4):619-31, iv-v. PMID 11567922
- [Background] James G, Doe T. The craniocervical flexion test: intra-tester reliability in asymptomatic subjects. Physiother Res Int. 2010 Sep;15(3):144-9. doi: 10.1002/pri.456. PMID 20146239
- [Background] Jull G, Barrett C, Magee R, Ho P. Further clinical clarification of the muscle dysfunction in cervical headache. Cephalalgia. 1999 Apr;19(3):179-85. doi: 10.1046/j.1468-2982.1999.1903179.x. PMID 10234466
- [Background] Jull GA, Falla D, Vicenzino B, Hodges PW. The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Man Ther. 2009 Dec;14(6):696-701. doi: 10.1016/j.math.2009.05.004. Epub 2009 Jul 25. PMID 19632880
- [Background] Jull GA, O'Leary SP, Falla DL. Clinical assessment of the deep cervical flexor muscles: the craniocervical flexion test. J Manipulative Physiol Ther. 2008 Sep;31(7):525-33. doi: 10.1016/j.jmpt.2008.08.003. PMID 18804003
- [Background] Juul T, Langberg H, Enoch F, Sogaard K. The intra- and inter-rater reliability of five clinical muscle performance tests in patients with and without neck pain. BMC Musculoskelet Disord. 2013 Dec 3;14:339. doi: 10.1186/1471-2474-14-339. PMID 24299621
- [Background] Kaufman-Cohen Y, Ratzon NZ. Correlation between risk factors and musculoskeletal disorders among classical musicians. Occup Med (Lond). 2011 Mar;61(2):90-5. doi: 10.1093/occmed/kqq196. Epub 2011 Jan 26. PMID 21273187
- [Background] Kibler WB, McMullen J. Scapular dyskinesis and its relation to shoulder pain. J Am Acad Orthop Surg. 2003 Mar-Apr;11(2):142-51. doi: 10.5435/00124635-200303000-00008. PMID 12670140
- [Background] Kibler WB, Sciascia A. Current concepts: scapular dyskinesis. Br J Sports Med. 2010 Apr;44(5):300-5. doi: 10.1136/bjsm.2009.058834. Epub 2009 Dec 8. PMID 19996329
- [Background] Kibler WB, Sciascia A, Wilkes T. Scapular dyskinesis and its relation to shoulder injury. J Am Acad Orthop Surg. 2012 Jun;20(6):364-72. doi: 10.5435/JAAOS-20-06-364. PMID 22661566
- [Background] Kibler WB, Sciascia AD. Introduction to the Second International Conference on Scapular Dyskinesis in Shoulder Injury--the 'Scapular Summit' Report of 2013. Br J Sports Med. 2013 Sep;47(14):874. doi: 10.1136/bjsports-2013-092424. Epub 2013 Apr 11. No abstract available. PMID 23580419
- [Background] Kibler WB, Ludewig PM, McClure PW, Michener LA, Bak K, Sciascia AD. Clinical implications of scapular dyskinesis in shoulder injury: the 2013 consensus statement from the 'Scapular Summit'. Br J Sports Med. 2013 Sep;47(14):877-85. doi: 10.1136/bjsports-2013-092425. Epub 2013 Apr 11. PMID 23580420
- [Background] Leaver R, Harris EC, Palmer KT. Musculoskeletal pain in elite professional musicians from British symphony orchestras. Occup Med (Lond). 2011 Dec;61(8):549-55. doi: 10.1093/occmed/kqr129. Epub 2011 Oct 14. PMID 22003061
- [Background] Lexell JE, Downham DY. How to assess the reliability of measurements in rehabilitation. Am J Phys Med Rehabil. 2005 Sep;84(9):719-23. doi: 10.1097/01.phm.0000176452.17771.20. PMID 16141752
- [Background] Mehrparvar AH, Mostaghaci M, Gerami RF. Musculoskeletal disorders among Iranian instrumentalists. Med Probl Perform Art. 2012 Dec;27(4):193-6. PMID 23247875
- [Background] McClure P, Tate AR, Kareha S, Irwin D, Zlupko E. A clinical method for identifying scapular dyskinesis, part 1: reliability. J Athl Train. 2009 Mar-Apr;44(2):160-4. doi: 10.4085/1062-6050-44.2.160. PMID 19295960
- [Background] O'Leary S, Falla D, Jull G. The relationship between superficial muscle activity during the cranio-cervical flexion test and clinical features in patients with chronic neck pain. Man Ther. 2011 Oct;16(5):452-5. doi: 10.1016/j.math.2011.02.008. Epub 2011 Mar 10. PMID 21396876
- [Background] Olson LE, Millar AL, Dunker J, Hicks J, Glanz D. Reliability of a clinical test for deep cervical flexor endurance. J Manipulative Physiol Ther. 2006 Feb;29(2):134-8. doi: 10.1016/j.jmpt.2005.12.009. PMID 16461172
- [Background] Paarup HM, Baelum J, Holm JW, Manniche C, Wedderkopp N. Prevalence and consequences of musculoskeletal symptoms in symphony orchestra musicians vary by gender: a cross-sectional study. BMC Musculoskelet Disord. 2011 Oct 7;12:223. doi: 10.1186/1471-2474-12-223. PMID 21978278
- [Background] Quarrier NF. Performing arts medicine: the musical athlete. J Orthop Sports Phys Ther. 1993 Feb;17(2):90-5. doi: 10.2519/jospt.1993.17.2.90. PMID 8467339
- [Background] Ranelli S, Straker L, Smith A. Playing-related musculoskeletal problems in children learning instrumental music: the association between problem location and gender, age, and music exposure factors. Med Probl Perform Art. 2011 Sep;26(3):123-39. PMID 21987067
- [Background] Sim J, Wright CC. The kappa statistic in reliability studies: use, interpretation, and sample size requirements. Phys Ther. 2005 Mar;85(3):257-68. PMID 15733050
- [Background] Steinmetz A, Moller H, Seidel W, Rigotti T. Playing-related musculoskeletal disorders in music students-associated musculoskeletal signs. Eur J Phys Rehabil Med. 2012 Dec;48(4):625-33. Epub 2012 Nov 9. PMID 23138678
- [Background] Steinmetz A, Seidel W, Muche B. Impairment of postural stabilization systems in musicians with playing-related musculoskeletal disorders. J Manipulative Physiol Ther. 2010 Oct;33(8):603-11. doi: 10.1016/j.jmpt.2010.08.006. Epub 2010 Oct 12. PMID 21036282
- [Background] Struyf F, Nijs J, Mollekens S, Jeurissen I, Truijen S, Mottram S, Meeusen R. Scapular-focused treatment in patients with shoulder impingement syndrome: a randomized clinical trial. Clin Rheumatol. 2013 Jan;32(1):73-85. doi: 10.1007/s10067-012-2093-2. Epub 2012 Oct 2. PMID 23053685
- [Background] Wilke C, Priebus J, Biallas B, Frobose I. Motor activity as a way of preventing musculoskeletal problems in string musicians. Med Probl Perform Art. 2011 Mar;26(1):24-9. PMID 21442133
- [Background] Zaza C, Farewell VT. Musicians' playing-related musculoskeletal disorders: an examination of risk factors. Am J Ind Med. 1997 Sep;32(3):292-300. doi: 10.1002/(sici)1097-0274(199709)32:33.0.co;2-q. PMID 9219660
- [Background] Zaza C. Playing-related musculoskeletal disorders in musicians: a systematic review of incidence and prevalence. CMAJ. 1998 Apr 21;158(8):1019-25. PMID 9580730
- [Background] Kava K, Larson C, Stiller C, Maher S. Trunk endurance exercise and the effect on instrumental performance: a preliminary study comparing pilates exercise and a trunk and proximal upper extremity endurance exercise program. Music Performance Research. Royal Northern College of Music. 2010;3(1):1-30
- [Derived] Silva FM, Brismee JM, Sizer PS, Hooper TL, Robinson GE, Diamond AB. Musicians injuries: Upper quarter motor control deficits in musicians with prolonged symptoms - A case-control study. Musculoskelet Sci Pract. 2018 Aug;36:54-60. doi: 10.1016/j.msksp.2018.04.006. Epub 2018 Apr 27. PMID 29738929